CLINICAL TRIAL: NCT01690247
Title: Human Umbilical Cord Mesenchymal Stem Cell Induce Liver Allografts Tolerance
Brief Title: Human Mesenchymal Stem Cells Induce Liver Transplant Tolerance
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Principal Investigator, Fu-Sheng Wang, Research Center for Biotherapy, Beijing 302 Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Beijing302-008
Record Dates: First submitted 2012-09-19; First posted 2012-09-21 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Evidence of Liver Transplantation
Keywords: mesenchymal stem cells; liver transplantation; clinical trial; rejection
MeSH Terms: conditions — Rejection, Psychology | interventions — Congresses as Topic; Immunosuppressive Agents; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional plus UC-MSC (Experimental): Participants will receive conventional treatment plus a dose of UC-MSC from day 0 through the week 12 study visit. Participants will then be followed until the week 48 study visit
  Interventions: Drug: Conventional plus UC-MSC
- Conventional plus placebo (Placebo Comparator): Participants will receive conventional plus placebo treatment from day 0 through the week 12 study visit. Participants will then be followed until the week 48 study visit.
  Interventions: Drug: Conventional plus placebo

INTERVENTIONS:
Drug: Conventional plus UC-MSC — Received conventional treatment and taken i.v., once per 4 week, at a dose of 1×106 UC-MSC/kg body weight for 12 weeks.
  Other Names: Immunosuppressive agents plus umbilical cord stem cells
  Arms: Conventional plus UC-MSC
Drug: Conventional plus placebo — Received conventional treatment and taken i.v., once per 4 week, at 50 ml saline for 12 weeks.
  Other Names: Immunosuppressive agents plus saline
  Arms: Conventional plus placebo

SUMMARY:
Liver transplantation is the only lifesaving intervention for patients with end-stage liver diseases. Despite the ability of current immunosuppressive agents to reduce the incidence of acute rejection, the rate of acute rejection reaches to 20-50% after liver transplantation. Furthermore, the long-term toxicity associated with current regimens for liver transplant recipients now is increasingly being perceived as an unmet clinical need. Mesenchymal stem cells (MSC) appeared to be effective in regulating the invoked immune response in setting such as tissue injury, transplantation, and autoimmunity, and have been used successfully to treat graft versus host disease and show immune modulation function both in vitro and in vivo and may help in repairing damaged tissue(s). Here, we evaluate umbilical cord derived MSC (UC-MSC) as an alternative immunosuppressive agents for liver transplanted patients, and examine if UC-MSC could improve the recovery of liver function.

DETAILED DESCRIPTION:
Liver transplantation is the only lifesaving intervention for patients with end-stage liver diseases. The current immunosuppressive agents reduce the incidence of acute cellular rejection; however, the rate of acute rejection reaches to 20-50% after liver transplantation. Furthermore, the long-term side effects of these regimens now has become a major challenge for liver transplant recipients and is increasingly being perceived as an unmet clinical need, for example, increases in the incidence of bacterial, viral infections, nephrotoxicity with chronic renal impairment, de novo diabetes mellitus, hyperlipidemia, arterial hypertension, cardiovascular disease, osteoporosis, neurotoxicity, hematological toxicity.

Mesenchymal stem cells (MSC) appeared to be effective in regulating the invoked immune response in setting such as tissue injury, transplantation, and autoimmunity, and have been used successfully to treat graft versus host disease and show immune modulation function both in vitro and in vivo and may help in repairing damaged tissue(s). Current clinical trails demonstrated that the use of autologous bone marrow MSC (BM-MSC) for renal transplanted patients resulted in lower incidence of acute rejection, decreased risk of opportunistic infection, and better estimated renal function. Compared with BM-MSC, umbilical cord derived MSC (UC-MSC) may be the better choice for clinical application. One main reason is that the collection of BM-MSC from liver transplanted patients would be harmful for the patients. Moreover, the proliferative abilities of BM-MSC from patients with liver disease are deficient, whereas, UC-MSC can be obtained from discarded umbilical cords and can be produced on a larger scale. Our and other studies reported that the infusion of human UC-MSC are feasible and can improve liver function of liver fibrosis and liver failure.

The purpose of this study is to learn whether and how UC-MSC can improve the conditions in liver transplanted patients. This study will also look at how well UC-MSC is tolerated and its safety in liver transplanted patients.

Participants in the study will be randomly assigned to one of two treatment arms:

Arm A: Participants will receive 12 weeks of standard regular immunosuppressive agents plus UC-MSC treatment. Arm B: Participants will receive 12 weeks of standard regular immunosuppressive agents plus placebo. UC-MSC will be prepared according to standard procedures and is collected in plastic bags containing anti coagulant. MSCs are given via i.v. under sonography monitoring. After UC-MSC transfusion, patients are followed up at week 4, 8, 12, 24, 36 and 48, and the evaluation of liver function recovery was performed.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Patients must be between the ages of 18 and 70 years and meet the criteria for liver transplantation.
3. Patient is receiving the first liver transplant.
4. Patient is receiving a liver transplant only.
5. Negative pregnancy test (female patients in fertile age).
6. Willing to comply with the study visits.

Exclusion Criteria:

1. Previously received or is receiving an organ transplant other than a liver.
2. Vital organs failure (Cardiac, Renal or Respiratory, et al).
3. Currently receiving an investigational drug or received an investigational drug within 30 days prior to transplant.
4. Currently receiving any immunosuppressive agent.
5. Clinically active bacterial, fungal, viral or parasitic infection.
6. Pregnant or lactating women.
7. Other candidates who are judged to be not applicable to this study by investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-02; Primary Completion 2014-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of acute rejection and early liver function recovery | 48 weeks

SECONDARY OUTCOMES:
Patient and graft survival, and prevalence of adverse events | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Sheng Wang, PHD, Principal Investigator — Beijing 302 Hospital
Locations (1):
- Beijing 302 Hospital, Beijing, China

REFERENCES:
- [Result] Tan J, Wu W, Xu X, Liao L, Zheng F, Messinger S, Sun X, Chen J, Yang S, Cai J, Gao X, Pileggi A, Ricordi C. Induction therapy with autologous mesenchymal stem cells in living-related kidney transplants: a randomized controlled trial. JAMA. 2012 Mar 21;307(11):1169-77. doi: 10.1001/jama.2012.316. PMID 22436957
- [Result] Perico N, Casiraghi F, Introna M, Gotti E, Todeschini M, Cavinato RA, Capelli C, Rambaldi A, Cassis P, Rizzo P, Cortinovis M, Marasa M, Golay J, Noris M, Remuzzi G. Autologous mesenchymal stromal cells and kidney transplantation: a pilot study of safety and clinical feasibility. Clin J Am Soc Nephrol. 2011 Feb;6(2):412-22. doi: 10.2215/CJN.04950610. Epub 2010 Oct 7. PMID 20930086
- [Result] Le Blanc K, Frassoni F, Ball L, Locatelli F, Roelofs H, Lewis I, Lanino E, Sundberg B, Bernardo ME, Remberger M, Dini G, Egeler RM, Bacigalupo A, Fibbe W, Ringden O; Developmental Committee of the European Group for Blood and Marrow Transplantation. Mesenchymal stem cells for treatment of steroid-resistant, severe, acute graft-versus-host disease: a phase II study. Lancet. 2008 May 10;371(9624):1579-86. doi: 10.1016/S0140-6736(08)60690-X. PMID 18468541
- [Result] Shi M, Liu ZW, Wang FS. Immunomodulatory properties and therapeutic application of mesenchymal stem cells. Clin Exp Immunol. 2011 Apr;164(1):1-8. doi: 10.1111/j.1365-2249.2011.04327.x. Epub 2011 Feb 24. PMID 21352202
- [Result] Zhang Z, Lin H, Shi M, Xu R, Fu J, Lv J, Chen L, Lv S, Li Y, Yu S, Geng H, Jin L, Lau GK, Wang FS. Human umbilical cord mesenchymal stem cells improve liver function and ascites in decompensated liver cirrhosis patients. J Gastroenterol Hepatol. 2012 Mar;27 Suppl 2:112-20. doi: 10.1111/j.1440-1746.2011.07024.x. PMID 22320928